CLINICAL TRIAL: NCT04339127
Title: Study of 12 Cases of Autoimmune Encephalitis With Anti-NMDA Receptor Antibodies Following Herpetic Encephalitis and Review of the Literature
Brief Title: Autoimmune Encephalitis With Anti-NMDA Receptor Antibodies Following Herpetic Encephalitis
Acronym: NMDARE-HSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: NMDARE-HSE
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Autoimmune Encephalitis; Anti NMDA Receptor Encephalitis; Herpetic Encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System; Anti-N-Methyl-D-Aspartate Receptor Encephalitis; Encephalitis, Herpes Simplex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort NMDARE-HSE: Patients developing clinical autoimmune encephalitis with anti-NMDA antibodies after a herpetic encephalitis, managed by the National Reference Center for Paraneoplastic Syndromes and Autoimmune Encephalitis at the Neurological Hospital of Bron.
  Interventions: Other: Description and analysis

INTERVENTIONS:
Other: Description and analysis — Retrospective, non-interventional study, using clinical, biological, radiological and therapeutic data collected during the initial diagnosis and follow-up.

SUMMARY:
Herpes Simplex Virus encephalitis is the most common infectious encephalitis, with an estimated annual incidence of 1 / 250,000 to 1 / 500,000 in industrialized countries. Despite a widely used antiviral treatment, the prognosis remains poor with a mortality of 5 to 20% and a considerable morbidity rate.

One of the contributing factors of bad prognosis is the development of encephalitis mediated by autoantibodies, most often directed against NMDA receptors, in the weeks following viral encephalitis.

The description of this pathology is recent, the pathophysiology of this process remains poorly understood, and the management of these patients is not yet codified.

ELIGIBILITY:
Inclusion Criteria:

* Clinical autoimmune encephalitis with anti-NMDA antibodies and documented by CBA in the CSF
* After a herpetic encephalitis documented by a positive viral PCR for HSV in the CSF
* Without age limit

Exclusion Criteria- No respect of inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 12 patients diagnosed between January 2014 and January 2020
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Details of clinical, biological, imaging, therapeutic characteristics and patient's evolution. | at 6 and 12 months
  Retrospective collection of clinical, diagnostic and therapeutic data, evolution at 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Honnorat, Study Director — National Reference Center of autoimmune encephalitis
Locations (1):
- Hospice Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No